CLINICAL TRIAL: NCT02569411
Title: Contacting Authors to Retrieve Individual Patient Data: Protocol for a Randomized Controlled Trial
Brief Title: Contacting Authors to Retrieve Individual Patient Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Andrea Tricco, Dr., Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-240c
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Response Rates

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- No Incentive (No Intervention): Those allocated to the control group will be contacted by email, mail, and phone, but will not receive a financial incentive
- Incentive (Experimental): Those allocated to the intervention group will be contacted by email, mail, and phone, and will be asked to provide the IPD from their RCT and they will be given a financial incentive.
  Interventions: Other: Financial Incentive

INTERVENTIONS:
Other: Financial Incentive — money
  Arms: Incentive

SUMMARY:
The objective of this study is to examine the impact of incentivizing authors of RCTs that are eligible for a systematic review and meta-analysis, versus usual contact strategies to obtain original IPD

ELIGIBILITY:
Inclusion Criteria:

* Corresponding authors of RCTs included in our previous and updated systematic reviews

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

REFERENCES:
- [Derived] Veroniki AA, Ashoor HM, Le SPC, Rios P, Stewart LA, Clarke M, Mavridis D, Straus SE, Tricco AC. Retrieval of individual patient data depended on study characteristics: a randomized controlled trial. J Clin Epidemiol. 2019 Sep;113:176-188. doi: 10.1016/j.jclinepi.2019.05.031. Epub 2019 May 30. PMID 31153977
- [Derived] Veroniki AA, Straus SE, Ashoor H, Stewart LA, Clarke M, Tricco AC. Contacting authors to retrieve individual patient data: study protocol for a randomized controlled trial. Trials. 2016 Mar 15;17(1):138. doi: 10.1186/s13063-016-1238-z. PMID 26975720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Authors identified in randomized controlled trials that were eligible for inclusion in two systematic review and network meta-analysis papers.
Pre-assignment Details: Authors whose contact information was unidentifiable were excluded.
Groups:
- No Incentive (Control): Those allocated to the control group will be contacted using the same approaches as the intervention arm for their participation to share individual patient data of their study. No financial incentive is provided.
- Financial Incentive (Intervention): Those allocated to the intervention group will be contacted by email, mail, and phone to share individual patient data from their study. They will be given a financial incentive (an offer of a $100 CAD gift card at first contact (or equivalent amount in the author's relevant currency) for their participation to share individual patient data of their study).
Period: Overall Study
Arm/Group | No Incentive (Control) | Financial Incentive (Intervention)
Started (Authors were contacted in either arm to share complete individual patient data during the study) | 65 | 64
Completed (None of the authors contacted in either arm shared complete individual patient data during the study) | 0 | 0
Not Completed | 65 | 64

BASELINE CHARACTERISTICS:
Population: Baseline data not collected on any participants
Groups:
- Total: Total of all reporting groups
Arm/Group | No Incentive | Incentive | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Customized
Sex/Gender, Customized
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Authors Who Provided Complete IPD
Description: We contacted authors of eligible studies from June 2016 to October 2016. Authors were first contacted in June 2016, where we sent: a) an email requesting their IPD, b) email reminders (4 in total) at 2, 6, 10, and 14-week intervals after the initial email, c) reminders by post in week 7, and d) reminders via telephone in week 15.
Time Frame: June 2016 - October 2016
Population: None of the authors in either arm shared individual patient data from their study.
Measure: Count of Participants; unit: Participants
Arm/Group | No Incentive (Control) | Financial Incentive (Intervention)
Number analyzed (Participants) | 65 | 64
Participants | 0 | 0

2. Secondary Outcome: Time Taken to Obtain the IPD Between Initial Request and Authors' Provision
Description: as for outcome 1
Time Frame: June 2016 - October 2016
Population: None of the authors in either arm shared individual patient data from their study therefore no data collected for this Outcome Measure.
Arm/Group | No Incentive (Control) | Financial Incentive (Intervention)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Completeness of the IPD Received
Description: as for outcome 1
Time Frame: June 2016 - October 2016
Population: as for outcome 2
Arm/Group | No Incentive (Control) | Financial Incentive (Intervention)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable. This study is non-clinical and so adverse event data was not collected.
Description: Not applicable. This study is non-clinical and so adverse event data was not collected.
Arm/Group | No Incentive (Control) | Financial Incentive (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT02569411/Prot_SAP_000.pdf